CLINICAL TRIAL: NCT04810429
Title: Comparison of Temporomandibular Joint Arthroscopy With Botulinum Toxin Injection Versus Placebo: a Randomized Clinical Trial
Brief Title: Comparison of Temporomandibular Joint Arthroscopy With Botulinum Toxin Injection Versus Placebo
Acronym: ARTHROBTX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Portugues da Face (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Eudrac: 2020-005610-18
Record Dates: First submitted 2021-03-11; First posted 2021-03-23 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-06

CONDITIONS: Temporomandibular Joint Disorders
Keywords: IncobotulinumoxinA; Temporomandibular Joint Disorder; Temporomandibular Joint arthroscopy; Randomized clinical trial
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Intervention Model Description: For this randomized clinical trial an appropriate number of sealed envelopes will be prepared: 15 for placebo and 15 for the treated group. Patients with inclusion criteria will be seen in an orofacial pain session and assessed for pain using the VAS scale, by scoring the degree of pain between 0 (absence of pain) and 10 (maximum pain). Then the patients are proposed for TMJ arthroscopy. The nurse enters the room with the patient and asks to the patient to choose an envelope. In this moment, the envelope is placed on a table and the patient writes his name. The nurse accompanies the patient to the doctor's office. Alone, the nurse opens the envelope and sees the code and the indication of PLACEBO or BTXA. Then, she will prepare in her room, isolated from the whole team, 2 syringes. She will put the envelope in a bag and deliver a tray with 2 syringes for treatment and a code to identify the patient in the treatment room. The doctor injects the syringes according to the protocol.
Who Masked: Investigator
Masking Description: atients with inclusion criteria will be seen in an orofacial pain session and assessed for pain using the VAS scale, by scoring the degree of pain between 0 (absence of pain) and 10 (maximum pain). Then the patients are proposed for TMJ arthroscopy. The nurse enters the room with the patient and asks to the patient to choose an envelope. In this moment, the envelope is placed on a table and the patient writes his name. The nurse accompanies the patient to the doctor's office. Alone, the nurse opens the envelope and sees the code and the indication of PLACEBO or BTXA. Then, she will prepare in her room, isolated from the whole team, 2 syringes. She will put the envelope in a bag and deliver a tray with 2 syringes for treatment and a code to identify the patient in the treatment room. The doctor injects the syringes according to the protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): TMJ arthroscopy and Saline solution NaCl 0,9% in 2 syringes with 1 ml each. Injected in Right Masseter (0.5ml), Left Masseter (0.5ml), Right Temporalis (0.5ml) and Left Temporalis (0.5ml).
  Interventions: Procedure: TMJ surgical arthroscopy
- IncobotulinumoxinA (Active Comparator): TMJ arthroscopy and Dose of IncobotulinumoxinA to be injected 100 U distributed in 2 syringes with 1 ml each: 25U (0.5ml) in Right Masseter / 25U (0.5ml) in Left Masseter / 25U (0.5ml) in Right Temporalis / 25U in Left Temporalis.
  Interventions: Drug: Incobotulinumoxin A; Procedure: TMJ surgical arthroscopy

INTERVENTIONS:
Drug: Incobotulinumoxin A — XEOMIN® (incobotulinumtoxinA) is an approved medication that inhibits the release of acetylcholine and muscle blockage. Xeomin is indicated for the symptomatic treatment of blepharospasm and hemifacial spasm, cervical dystonia of a predominantly rotational type (spasmodic torticollis), spasticity of the upper limbs and chronic sialorrhea due to neurological changes. Xeomin comes as a white powder for solution for injection. When dissolved Xeomin is a clear, colorless solution that does not contain particles. Xeomin is reconstituted before use with sterile sodium chloride 9 mg / ml (0.9%) solution, without preservatives, for injections.
  The active substance is Clostridium botulinum type A neurotoxin (150 kD), without complexing proteins. The other components are human albumin and sucrose.
  Arms: IncobotulinumoxinA
Procedure: TMJ surgical arthroscopy — TMJ arthroscopy is a minimal invasive surgical technique for different types of temporomandibular joint (TMJ) internal derangements. Besides the acceptable outcomes of TMJ arthroscopy, the authors believe that adding to this treatment a single injection of BTXA into the temporalis and masseter muscles could reduce joint loading, improving TMJ arthroscopic results.

SUMMARY:
There are several studies that have considered Botulinum toxin A (BoNT-A) injections are effective in treating symptoms for Temporomandibular Joint (TMJ) disorders. BoNT-A injections improve the hyper-tonicity of mandibular muscles and its consequent joint load reduction. Also injections of BoNT-A, for patients with articular disc displacement, resulted in pain relief and return of the normal movements of the mandible. The main goal of this study is to test the beneficial impact of BoNT-A injections in the masticatory muscles of patients submitted to TMJ surgical arthroscopy.

DETAILED DESCRIPTION:
Study Objective:

To investigate the potential performance of incobotulinumtoxin-A (BTXA) in patients submitted to TMJ surgical arthroscopy. Besides the acceptable good outcomes of TMJ arthroscopy, the authors believe that using a single injection of BTXA into the temporalis and masseter muscles could reduce joint loading and pain, improving TMJ arthroscopy results.

The proposed explanation for this study:

TMJ arthroscopy is a minimal invasive surgical technique for different types of temporomandibular joint (TMJ) internal derangements. Besides the acceptable outcomes of TMJ arthroscopy, the authors believe that adding to this treatment a single injection of BTXA into the temporalis and masseter muscles could reduce joint loading, improving TMJ arthroscopic results.

ELIGIBILITY:
Inclusion Criteria:

* Patients with TMJ with indication for arthroscopy
* Age between 12-60 years old
* Minimum level of pain for inclusion should be 5/10 (on a 0-10 VAS scale)

Exclusion Criteria:

* Previous treatment to TMD
* Previous use of facial Botulinum Toxin
* Any contraindication for the use of BTXA according to XEOMIN SmPC

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
VAS score | 5 weeks after injection and TMJ arthroscopy
  Improvement in TMJ pain: measured by the patient using a Visual Analogue scale (VAS), with a range from 0 to 10, with 0 being no pain and 10 having maximum unbearable pain. VAS score will be measured every week before surgery and in the fifth week after surgery.

SECONDARY OUTCOMES:
Palpable joint click | 5 weeks after injection and TMJ arthroscopy
  Yes or No
Diet consistency tolerated | 5 weeks after injection and TMJ arthroscopy
  regular diet, basic diet, liquid diet
Muscle Tenderness | 5 weeks after injection and TMJ arthroscopy
  Masseter muscle, temporalis muscle, temporalis tendon, and lateral capsule of the TMJ) - Muscle sensitivity scale (0-3)
Maximum Mouth Opening | 5 weeks after injection and TMJ arthroscopy
  in cm
GICS | 5 weeks after injection and TMJ arthroscopy
  Global Impression of change by the subject

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Português da Face, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Yes
A study Protocol and clinical study report will be avaiable in the end of the study.
Supporting Information: Study Protocol, CSR
Time Frame: At the moment it is not possible to predict